CLINICAL TRIAL: NCT05301296
Title: Evaluating of Clinical Early Detection of Breast Cancer in Trivandrum District, India
Brief Title: Trivandrum Breast Cancer Screening Trial
Acronym: TBCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Regional Cancer Centre, Trivandrum, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IEC 05-05
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Detection of Cancer

STUDY DESIGN:
Intervention Model Description: The control group received standard of care while the intervention group received 3 rounds of screening with clinical breast examination, each 3 years apart. After the 3 rounds of screening, the participants were followed up for an additional 4 years to accrue information on breast cancer incidence and mortality, and the vital status.
Masking Description: Cancer registry staff members blinded to study group assignments collected data on the date of diagnosis, stage, treatment and follow-up details of breast cancer patients by visiting hospitals and laboratories where breast cancer cases are diagnosed and treated. The cause of death was assessed by two independent experts blinded to group allocation after evaluation of data from hospital records, death certificates, house visits and interviews of relatives and friends.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Standard of Care.
- Intervention Arm (Active Comparator): Clinical examination of the breast for early detection of Cancer.
  Interventions: Diagnostic Test: Clinical examination of the breast for early detection of Cancer

INTERVENTIONS:
Diagnostic Test: Clinical examination of the breast for early detection of Cancer — Participants were invited for 3 rounds of clinical breast examination, conducted 3-years apart. Screening was conducted by health workers trained to perform clinical breast examination for early detection of cancer. Women with abnormal referable lesions underwent CBE by a trained clinician and those women with a confirmed breast lump or any other breast abnormality warranting further investigations were evaluated by triple-testing involving expert physical examination, diagnostic mammography with or without ultrasonography and fine needle aspiration cytology (FNAC) or core biopsy or excision biopsy. Those with confirmed breast cancer were referred for appropriate treatment with surgery, radiotherapy, and/or chemotherapy.
  Arms: Intervention Arm

SUMMARY:
Cluster-randomized controlled trial in Trivandrum district, Kerala, India to evaluate the effect of triennial screening for breast cancer using clinical breast examination on breast cancer mortality.

DETAILED DESCRIPTION:
The study population consisted of 274 administrative regions (clusters) in Trivandrum district, Kerala, southern Indian. 133 clusters were randomly assigned to the intervention arm (3 rounds of clinical breast examination conducted 3 years apart) and were compared to the remaining 141 clusters assigned to a control arm that received standard of care. The eligibility criteria were all healthy subjects aged 30 to 69, without a personal history of breast cancer. Informed consent was signed by each participant. The intervention arm consisted of 55,843 participants and the control group consisted of 59,447 participants.

ELIGIBILITY:
Inclusion Criteria:

* Residing in 274 study clusters in Trivandrum City, Kerala

Exclusion Criteria:

* Diagnosis with breast cancer prior to study
* Bedridden subjects
* Subjects suffering from open tuberculosis or other debilitating diseases

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115290 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Death Rate | 14 years
  Information on all deaths were collected from the municipal and district death registers, hospital medical records, death records of churches and mosques, hospital visits by the population cancer registry staff and by project health workers. Cancer cases were coded by the ICD-O 3rd edition codes and cause of death was coded using ICD-10 by the registry and project staff blinded to study group allocation. Deaths were attributed to breast cancer if the patient had histologically or clinically confirmed breast cancer, lymph nodes or distant metastasis at the time of death or had died due to complications of breast cancer treatment.
Breast Cancer Incidence | 14 years
  Information on incident breast cancer cases were obtained from the Trivandrum population-based cancer registry, hospital cancer registry of the RCC and medical records departments of other hospitals treating breast cancer patients. Collection of information was blinded to study group assignment of cases. The staging of breast cancers was done according to the UICC TNM staging system.

CONTACTS AND LOCATIONS:
Overall Officials: Kunnambath Ramadas, MD. DNB. FAMS, PhD, Principal Investigator — Regional Cancer Centre, Trivandrum, India; Rengaswamy Sankaranarayanan, MD, Principal Investigator — International Agency for Research on Cancer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sankaranarayanan R, Ramadas K, Thara S, Muwonge R, Prabhakar J, Augustine P, Venugopal M, Anju G, Mathew BS. Clinical breast examination: preliminary results from a cluster randomized controlled trial in India. J Natl Cancer Inst. 2011 Oct 5;103(19):1476-80. doi: 10.1093/jnci/djr304. Epub 2011 Aug 23. PMID 21862730